CLINICAL TRIAL: NCT02096991
Title: Associations of Exposure to Bisphenol A With Blood Pressure and Epigenetic Change
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Yun-Chul Hong, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: BPA-CAN-1
Record Dates: First submitted 2014-02-02; First posted 2014-03-26 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — allergen Can f 2; Glass

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Glass (Active Comparator): consume beverage in glass first and cross over to other interventions
  Interventions: Other: Can 1; Other: Can 2; Other: Glass
- Can 1 (Experimental): consume one canned beverage and a glass bottled beverage first and cross over to other interventions
  Interventions: Other: Can 1; Other: Can 2; Other: Glass
- Can 2 (Experimental): Consume two canned beverage first and cross over to other interventions
  Interventions: Other: Can 1; Other: Can 2; Other: Glass

INTERVENTIONS:
Other: Can 1 — drink the beverage in a can and a glass bottle
Other: Can 2 — Consume two canned beverage
Other: Glass — consume two glass bottled beverage

SUMMARY:
* Bisphenol A(BPA) is an endocrine disrupting chemical, which mimics the action of estrogen.
* Previous studies reported that BPA exposure is associated with increased risk of cardiovascular diseases.
* Exposure to BPA occur mainly through oral route, and epoxy coating of canned food is one of the well established source.
* The investigators hypothesis is that increased BPA exposure from canned beverage would disrupt normal physiology in a short term.
* In the present trial the investigators are to investigate whether increased BPA exposure by consuming canned beverage actually affect cardiovascular indices and epigenetic feature.
* For this aim, the investigators will conduct a cross-over trial.

ELIGIBILITY:
Inclusion Criteria:

* Reside in Seoul
* Who provided Informed consent

Exclusion Criteria:

* Who has cancer
* Who has disease or disorder of liver, nervous system, endocrine system, cardiovascular system
* Who does not provieded informed consent

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-02; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | 2 hours after consuming beverage

SECONDARY OUTCOMES:
Percent DNA methylation | 2 hours after consuming the beverage
Heart Rate Variablility | 2 hours after consuming the beverage

CONTACTS AND LOCATIONS:
Overall Officials: Yun-Chul Hong, MD, PhD, Principal Investigator — Department of Preventive Medicine, College of Medicine, Seoul National University
Locations (1):
- Department of Preventive Medicine, College of Medicine, Seoul National University, Seoul, South Korea

REFERENCES:
- [Derived] Bae S, Hong YC. Exposure to bisphenol A from drinking canned beverages increases blood pressure: randomized crossover trial. Hypertension. 2015 Feb;65(2):313-9. doi: 10.1161/HYPERTENSIONAHA.114.04261. Epub 2014 Dec 8. PMID 25489056